CLINICAL TRIAL: NCT04228185
Title: Banded Sleeve Gastrectomy Improves Weight Loss Compared to Non-banded Sleeve: Mid-term Results From a Prospective Randomized Study
Brief Title: Banded Sleeve Gastrectomy Improves Weight Loss Compared to Non-banded Sleeve: Mid-term Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Stefano D'Ugo, Principal Investigator, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Banded_Sleeve
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Obesity, Morbid
Keywords: Sleeve gastrectomy; banded sleeve; obesity surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic banded sleeve gastrectomy (Experimental): Group undergoing banded sleeve
  Interventions: Procedure: sleeve gastrectomy
- Laparoscopic sleeve gastrectomy (Active Comparator): Group undergoing standard sleeve
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: sleeve gastrectomy — Comparison of banded and not-banded sleeve gastrectomy

SUMMARY:
Weight regain after Laparoscopic Sleeve Gastrectomy (LSG) is nowadays a growing concern. Sleeve dilatation and loss of food restriction is considered the main mechanism. The placement of a silicon ring around the gastric tube seems to give benefits in the short-term.

The Investigators evaluate the efficacy of banded sleeve gastrectomy compared to standard sleeve in the mid-term.

Fifty patients were randomized between LSG and Laparoscopic Banded Sleeve Gastrectomy (LBSG), and they underwent a mean follow-up of 4 years.

Patients' management was exactly the same, apart from the band placement. After surgery differences in weight loss, operative time, complication rate and mortality were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity
* Failure of medical treatment
* >18yrs; <60 yrs

Exclusion Criteria:

* Previous bariatric or GI surgery
* Psychiatric disease
* Pregnancy
* Contraindication to laparoscopy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
weight loss | from surgery to 4 years follow up
  comparison of weight loss between the two procedures

SECONDARY OUTCOMES:
Complications | from surgery to 4 years follow up
  Short and mid-term complications

CONTACTS AND LOCATIONS:
Overall Officials: Stefano D'Ugo, MD PhD, Principal Investigator — Tor Vergata University Hospital
Locations (1):
- Tor Vergata University Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gentileschi P, Bianciardi E, Siragusa L, Tognoni V, Benavoli D, D'Ugo S. Banded Sleeve Gastrectomy Improves Weight Loss Compared to Nonbanded Sleeve: Midterm Results from a Prospective Randomized Study. J Obes. 2020 May 28;2020:9792518. doi: 10.1155/2020/9792518. eCollection 2020. PMID 32566276